CLINICAL TRIAL: NCT04514276
Title: Inter- and Multidisciplinary, Cross-sectoral Feto-neonatal Pathway for High-risk Pregnant Women Because of Fetal Growth Restriction
Brief Title: Inter- and Multidisciplinary, Cross-sectoral Feto-neonatal Pathway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Jena University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FetoNeonatPfad
Record Dates: First submitted 2020-06-22; First posted 2020-08-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pre-Eclampsia; Intrauterine Growth Restriction; Maternal Care for Known or Suspected Poor Fetal Growth
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- consecutive fetoneonatal healthcare (Experimental): inclusion criteria: pregnant woman having higher risk of early fetal growth restriction, preeclempsia living in studyregion (east-Saxony or east Thuringia) the fetoneonatal pathway consists of four consecutive parts: (1) early perceiving of pregnant women with higher risks for early fetal growth restrictions via color Doppler sonography, fetal biometry, haemogram check (currently additional screenings) (2) structured care of the high risk women who are pregnant (3) concerted neonatal health care (4) adapted paediatric aftercare, certain dates and responsible persons are scheduled.
  Interventions: Other: consecutive fetoneonatal healthcare pathway
- standard fetoneonatal healthcare (No Intervention): inclusion criteria: due to health insurance data by AOK PPLUS & ikk classics propsensityscorematched pregnant women living in west Saxony and Thuringia, being not part of the intervention group receiving standard health care.

INTERVENTIONS:
Other: consecutive fetoneonatal healthcare pathway — (1) early perceiving of pregnant women with higher risks for early fetal growth restrictions via color Doppler sonography, fetal biometry, haemogram check (currently additional screenings) (2) structured care of the high risk women who are pregnant (3) concerted neonatal health care (4) adapted paediatric aftercare, certain dates and responsible persons are scheduled.
  Arms: consecutive fetoneonatal healthcare

SUMMARY:
Due to the fetoneonatal pathway it is possible to identify pregnant women with an increased risk of fetal growth restriction or pre-eclampsia in early stages (from 10th week of pregnancy). Women whose pregnancy is considered high-risk receives risk-adapted prenatal treatment as well as certain treatments for their newborn and infant until 1 year of age. The tasks of all involved persons are defined by standard operating procedures (SOP)

DETAILED DESCRIPTION:
By implementing a preventive feto-neonatal pathway, healthcare for pregnant women with high risk of fetal growth restriction (FGR) or pre-eclampsia will be improved and, therefore the occurence of children's health problems may be prevented.The pathway allows healthcare to be structured, ross-sectoral, inter- and multidisciplinary in consideration of medical and psychosocial imensions. The feto-neonatal pathway transfers scientific findings, which already determine international routine care, in the project region into clinical routine care. The anamnestically increased risk for FGR or pre-eclampsia is validated by ultrasound and the identified high-risk pregnancy is attended risk-adapted from birth until the end of the first year of life of the child.As a result, the mothers' pregnancy-related risks (death, premature delivery, traumatic stress disorders) as well as risks for the child (prematurity and associated problems, childhood growth restriction with the risk of metabolic syndrome, developmental neurological problems) are reduced and the sustainability of the interventions is ensured in the long term through improved health competence of the families. The feto-neonatal pathway shows how highly specialised fetoneonatal care of high-risk pregnancies can be ensured while ensuring primary care in a health region, and offers the possibility of being extended to other indications.

ELIGIBILITY:
Inclusion Criteria:

* Female, minim. 10 weeks of pregnancy, maximum 36 weeks of pregnancy
* anamnestic risk of preeclempsia or fetal growth restriction
* being part of the project region

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnancy
Enrollment: 828 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of patients' safety: maternal pre-eclampsia rate | through study completion, an average of 1 year and 7 months
  self-designed questionnaire, health information
Evaluation of patients' safety: newborn's birthweight adjusted by gestational age | through study completion, an average of 1 year and 7 months
  self-designed questionnaire, health information
Evaluation of patients' safety: maternal morbidity | through study completion, an average of 1 year and 7 months
  self-designed questionnaire, health information
Evaluation of patients' safety: infantil morbidity | through study completion, an average of 1 year and 7 months
  self-designed questionnaire, health information
Evaluation of patients' safety: Quality of life | through study completion, an average of 1 year and 7 months
  Questionnaire: Quality of Life (Angermayer, Kilin & Matschinger, 2000)
Evaluation of patients' safety: attachment behavior | through study completion, an average of 1 year and 7 months
  Questionnaire: Postpartum Bonding Questionnaire (Reck et al., 2006)
Evaluation of patient's access to treatment and satisfaction | through study completion, an average of 1 year and 7 months
  self-designed questionnaire
claim of the health services | From admission to discharge, study inclusion to one year postpartum)
  based on self-designed questionnaires
prohibition of employment | From admission to discharge, study inclusion to one year postpartum)
  based on self-designed questionnaires
duration of unemployability | From admission to discharge, study inclusion to one year postpartum)
  based on self-designed questionnaires

SECONDARY OUTCOMES:
health economical evaluation | From admission to discharge, study inclusion to one year postpartum
  cost-benefit-analysis of patients' outcome in relation to supply costs based on secondary data provided by Health insurance funds
evaluation of ungoing processes during the fetoneontal health care pathway: target patients | From admission to discharge, study inclusion to one year postpartum
  based on secondary data provided by Health insurance funds
evaluation of ungoing processes during the fetoneontal health care pathway: effectiveness of fetoneonatal health care | From admission to discharge, study inclusion to one year postpartum
  based on secondary data provided by Health insurance funds
evaluation of ungoing processes during the fetoneontal health care pathway: participation of health care provider | From admission to discharge, study inclusion to one year postpartum
  based on secondary data provided by Health insurance funds
evaluation of ungoing processes during the fetoneontal health care pathway: implementation of participating employees | From admission to discharge, study inclusion to one year postpartum
  based on secondary data provided by Health insurance funds
evaluation of ungoing processes during the fetoneontal health care pathway: the pathway's maintenance being long term part of routine health care | From admission to discharge, study inclusion to one year postpartum
  based on secondary data provided by Health insurance funds

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rüdiger, Prof. Dr, Study Director — Technische Univeristät Dresden
Locations (2):
- Germany (2):
  - Medizinische Fakultät Dresden Klinik und Poliklinik für Kinder- und Jugendmedizin / Neonatologie & Pädiatrische Intensivmedizin, Dresden, Saxony
  - Universitätsklinikum Jena Klinik für Kinder- und Jugendmedizin, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No
data protection reasons

REFERENCES:
- [Derived] Epple F, Reichert J, Rudiger M, Birdir C, Mense L. Early psycho-social support of pregnant women at risk for preeclampsia and fetal intrauterine growth restriction. BMC Pregnancy Childbirth. 2025 Oct 27;25(1):1142. doi: 10.1186/s12884-025-08363-9. PMID 41146068
- See also: Medizinische Fakultät DresdenKlinik und Poliklinik für Kinder- und Jugendmedizin / Neonatologie & Pädiatrische Intensivmedizin — https://www.uniklinikum-dresden.de/de/das-klinikum/kliniken-polikliniken-institute/kik/bereiche/fachbereiche/neonatologie-its